CLINICAL TRIAL: NCT06449417
Title: Aurora's Impact on Mitigating Adverse Effects of Neoadjuvant Chemotherapy in Breast Cancer Patients in Chile's Metropolitan Region.
Brief Title: Aurora: a Human-centered Program for Breast Cancer Patients in Chile, Easing Neoadjuvant Chemotherapy's Effects
Acronym: Aurora
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 230126002
Record Dates: First submitted 2024-05-09; First posted 2024-06-10 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer
Keywords: Physical Activity; Quality of Life; Fatty Acids
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: This study is a mixed-methods Randomized Control Trial evaluating the impact of Aurora, a human-centered design, on breast cancer patients undergoing neoadjuvant chemotherapy in the Metropolitan Region of Chile. The study measures quantitative and qualitative variables over a 9-week intervention. The control group comprises patients without Aurora. The primary outcome is quality of life, with secondary outcomes including functional capacity and tumor progression. The study includes sociodemographic data extraction, baseline and intervention end measurements, and correlations between variables. The Aurora program integrates motivation, peer learning, and community support. The hypothesis is that Aurora enhances the biopsychosocial effects and mitigates adverse physical and biological consequences of breast cancer by promoting physical activity.
Who Masked: Outcomes Assessor
Masking Description: Blind statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aurora Training Group (Experimental): The experimental group will receive an online class of the benefits of physical activity for breast cancer patients, followed by the delivery of the human centered design intervention program.The Aurora kit is a plastic container including a resistance band, two 2 kg dumbbells, a therapeutic ball, an arm volume measurement tape, a hydration bottle for the patient, a leaflet with a guide of recommended exercises, and the logbook journal. The intervention lasts 9 weeks.
  Interventions: Behavioral: Experimental Aurora Training
- Control Group (No Intervention): The control group will receive an online class of the benefits of physical activity for breast cancer patients, followed by the delivery of the control kit.The control kit is a tote bag including a hydration bottle for the patient, and a logbook journal with blanc pages. The intervention lasts 9 weeks.

INTERVENTIONS:
Behavioral: Experimental Aurora Training — Patients will be asked to record their physical activity in the logbook every week, at the end of the intervention, each patient will have to dedicate a letter to another patient who will receive the same Aurora Kit.
  Arms: Aurora Training Group

SUMMARY:
Breast cancer is the most prevalent cancer worldwide and the leading cause of cancer death among women in Chile. The Aurora intervention program is designed to improve the quality of life and mitigate the physical consequences of breast cancer in patients undergoing neoadjuvant chemotherapy. It aims to promote physical activity through a human-centered design product system, incorporating elements of personal motivation, peer learning, and community engagement in alignment with the COM-B model.

In a 9-week randomized controlled trial, we will include 30 female patients under 70 years undergoing neoadjuvant therapy for breast cancer in the Metropolitan Region of Chile. Baseline and post-intervention measurements will assess biopsychosocial breast cancer effects through a questionnaire as well as adverse physical effects through functional capacity tests. Biological consequences will be evaluated through lipid profiling, inflammation biomarkers, and tumor progression. In addition, Aurora's patient perception of behavior change will be addressed by analyzing the patient's records in a journal. Moreover, the perceived value of Aurora's design attributes influencing behavior change will be studied through in-depth interviews.

Preliminary results describe Aurora's design process and indicate that it is well-received by patients, especially as its logbook is a valuable tool for self-reflection and progress tracking. The study anticipates the confirmation that significantly higher physical activity, improved quality of life, and enhanced functional capacity will be attained in the intervention group.

The Aurora intervention program represents a novel approach to support breast cancer patients undergoing chemotherapy, emphasizing physical activity, peer learning, and self-reflection. The integration of the behavior change COM-B model and a human-centered design provides a facilitating tool for tailored interventions for breast cancer patients' needs. Yet, the potential correlation between physical activity, fatty acid metabolism, and chemotherapy response necessitates further exploration.

The Aurora intervention program shows promise as a supportive tool for breast cancer patients undergoing neoadjuvant chemotherapy. Further research is imperative to evaluate the intervention's impact on patient outcomes, refine the design based on user feedback, and explore potential relationships among physical activity, fatty acid metabolism, and chemotherapy response.

DETAILED DESCRIPTION:
The research question of this project focuses on the quantitative and qualitative dimensions in health concerning temporality, specifically exploring and understanding health phenomena in a specific temporal context within the framework of the intervention with the Aurora human centered design product system therapeutic intervention program. The hypothesis is that the Aurora program significantly enhances the biopsychosocial breast cancer effects and mitigates breast cancer's adverse physical and biological consequences among women undergoing neoadjuvant chemotherapy in the Metropolitan Region of Chile by promoting physical activity. The main goal is to evaluate the impact of the Aurora product system therapeutic intervention program on enhancing the biopsychosocial effects and mitigating the adverse physical and biological consequences of breast cancer for women undergoing neoadjuvant chemotherapy in the Metropolitan Region of Chile by promoting physical activity.The specific objectives are:

i) Evaluate the impact of the Aurora human centered design product system therapeutic intervention program on Physical Activity levels (measured by intensity, time, and adherence) among women undergoing neoadjuvant chemotherapy in the Metropolitan Region of Chile by comparing the intervention and control groups at baseline and at the end of the program.

ii) Assess the effectiveness of the Aurora human centered design product system therapeutic intervention program in enhancing the biopsychosocial effects of breast cancer (measured by quality of life and patient´s perceptions) among women undergoing neoadjuvant chemotherapy in the Metropolitan Region of Chile by comparing the intervention and control groups at baseline and at the end of the program.

iii) Determine the extent to which the Aurora human centered design product system therapeutic intervention program mitigates the physical consequences of breast cancer (measured by functional capacity) among women undergoing neoadjuvant chemotherapy in the Metropolitan Region of Chile by comparing the intervention and control groups at baseline and at the end of the program.

iv) Examine the role of the Aurora human centered design product system therapeutic intervention program in reducing the biological consequences of breast cancer (measured by lipid profile LDL, HDL, and RBCm FA; inflammation by CRP and neutrophil to lymphocyte ratio; and tumor progression by residual cancer burden and pathological complete response) among women undergoing neoadjuvant chemotherapy in the Metropolitan Region of Chile by comparing the intervention and control groups at baseline and at the end of the program.The study program consists of four main phases: Week 0-4: Patients provide informed consent, and sociodemographic data, breast cancer subtype, and stages are collected. An online educational session is held, detailing physical activity advantages and outlining recommended exercise types, durations, and frequencies for breast cancer patients. Participants' availability is gathered to schedule an online assessment, which includes the quality of life questionnaire, functional capacity evaluations, and a dietary survey. Blood samples are drawn from routine tests in coordination with their neoadjuvant chemotherapy indication or schedule.

Week 4-13: Participants are randomized using minimization, considering each new participant's characteristics, such as age and cancer stage, which are determinant factors for physical activity adherence. Participants receive kits tailored to their assigned group, complete with instructions on using each item and what to document in the provided journal over the nine-week intervention period. Participants in the intervention group receive the Aurora human centered design product system, while those in the control group receive a kit with the same hydration bottle, measurement tape, a logbook journal with blank pages, and an electronic step count wristband, all packaged in an Aurora-branded tote bag. Weekly follow-ups ensure compliance with the protocol and record any adverse events.

Week 13-16: The research team coordinates the return of the kits. Participants in the intervention group return the container with all the sports equipment and the dedication letter to the next participant. The team confirms whether the participant wishes to keep the journal, and if so, each page is photographed for record-keeping before returning it to the participant. The participant also keeps the water bottle. In the control group, the same procedure is followed for the journal delivery, and participants keep the tote bag and the water bottle. They return the measurement tape and the pedometer. Prior to surgery, each patient undergoes routine blood sampling for testing, following the same procedure as at baseline.The experimental procedures involve determining physical activity levels, physical activity adherence, quality of life, and Aurora's perception. Physical activity levels are measured according to the number of exercise sessions reported on a weekly basis and their compliance with the reported minimum of 3 weekly sessions for breast cancer patients in Chile. The intervention group receives specially designed pages in their Aurora journal to register this information, whereas the control group has blank pages to record the data. Physical activity time is evaluated at baseline and at the end of the intervention with the International Physical Activity questionnaire in its short form. Physical activity intensity is measured using wrist pedometers provided by the Oncology physical therapy unit at Complejo Asistencial Dr. Sótero del Río. Quality of Life is assessed using the European Organization for Research and Treatment of Cancer (EORTC) QLQ-BR23 questionnaire at baseline and at the end of the intervention. To understand Aurora's perception, two methods are assessed at the end of the intervention: a thematic analysis of the Aurora journals and a system design evaluation. The reflections recorded in the Aurora logbook journal are transcribed and analyzed using an inductive thematic analysis following the COM-B constructs. The system design evaluation is conducted in online, in-depth, focused interview sessions with participants from the intervention group at the end of the last patient's cycle.

The method for extracting and measuring fatty acids (FA) involves drawing 5 ml of venous blood after a 12-hour fast, separating red blood cells, and extracting plasma membranes following a specific procedure. The FA from these membranes are then extracted using the Folch method, which uses a mixture of chloroform and methanol to extract lipids. The FA are derivatized to form fatty acid methyl esters (FAMEs) for analysis by gas chromatography to determine the fatty acid composition. Neutrophil and lymphocyte counts ratio (NLR) will be obtained from a complete blood count, and omega-3 (⍵-3) and omega-6 (⍵-6) PUFAs will be determined by extracting total lipids from red blood cells and total plasma. Residual cancer burden (RCB) and pathological complete response (pCR) will be calculated post-surgery based on data from electronic medical records to assess tumor progression.

The statistical analysis will be performed using R Studio, and the results will be analyzed under the intention-to-treat principle. Descriptive, inferential, and correlation analyses will be conducted, with statistical significance defined as p≤0.05. Descriptive statistics will present the results as the mean and standard deviation for continuous variables with a symmetrical distribution or as percentiles and range for continuous variables with an asymmetrical distribution. Inferential statistics will compare baseline characteristics and within-group and between-group differences using t-tests, Pearson´s chi-square tests, or non-parametric tests, respectively, for data distribution.

ELIGIBILITY:
Inclusion Criteria:

* Women under 70 years old
* Diagnosis of primary breast carcinoma,
* Indication for neoadjuvant chemotherapy
* Access to a safe physical space for performing PA
* Connection to the Internet
* Access to an electronic device for video conferencing

Exclusion Criteria:

* Stage IV cancer (non-curative)
* Medical contraindication to physical activity
* Self-report of physical activity participation equivalent to the current governmental physical exercise recommendation guide
* Body mass index lower than 18.5 kg/m2 or greater than 40 kg/m2.

Max Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Quality of Life Perception Score | 9 weeks
  To assess the effectiveness of the Aurora human centered design product system therapeutic intervention program in enhancing the biopsychosocial effects of breast cancer in women undergoing neoadjuvant chemotherapy in the metropolitan region of Chile, quality of life will be measured using the European Organization for Research and Treatment of Cancer (EORTC) questionnaire, the QLQ-BR23 (Quality of life questionnaire number 23 for breast cancer) is a module tailored to breast cancer patients, focusing on symptoms and issues relevant to this group.
  The EORTC QLQ-BR23 uses a 4-point Likert scale, where 1 represents "Not at all" and 4 represents "Very much." The scores are then transformed to a scale of 0 to 100, where higher scores indicate a higher level of symptoms or problems, and lower scores indicate a lower level of symptoms or problems.

SECONDARY OUTCOMES:
Patient Perception | 9 weeks
  Assess the effectiveness of the Aurora human centered design product system therapeutic intervention program in enhancing the biopsychosocial effects of breast cancer measured by by patient´s perceptions through a in depth interview, among women undergoing neoadjuvant chemotherapy in the metropolitan region of Chile by assessing the intervention group at the end of the program. Interviews will be transcribed and textual qualitative data will be analyzed to find emergent topics.
Lipid Profile | 9 weeks
  Examine the role of the Aurora human centered design product system therapeutic intervention program in reducing the biological consequences of breast cancer measured by lipid profile in plasma LDL, HDL, and RBCm fatty acids, among women undergoing neoadjuvant chemotherapy in the Metropolitan Region of Chile by comparing the intervention and control groups at baseline and at the end of the program.
Change on aerobic capacity measured with the Two-Minute Walk Test at baseline and at the end of the program. | 9 weeks
  The Two-Minute Walk Test is a simple performance-based test used to measure an individual's walking ability and functional capacity. In this test, the participant marches in place for two minutes, lifting their knees to a height midway between the patella (kneecap) and the iliac crest (hip bone). The number of times the right knee reaches this height is counted and recorded as the score. The variable measured is the number of repetitions completed within the 2-minutes timeframe, it is a quantitative discrete variable.
Change in arm volume measured with the 6 Measures Assessment of Arm Volume at baseline and at the end of the program. | 9 weeks
  This volume test is a method used to measure arm volume, which is an important indicator for detecting and monitoring lymphedema, a common complication after breast cancer treatment. The test involves taking circumferential measurements of the arm at 6 specific locations using a flexible tape measure. These circumferential measurements are then used to calculate the arm volume by modeling the arm segments as truncated cones and summing the volumes of the individual segments. The variable measured is the arm volume, which is a continuous quantitative variable expressed in units of volume in milliliters (mL).
Change in upper extremity strength measured with the 30-second elbow extension test at baseline and at the end of the program. | 9 weeks
  The 30-second elbow extension test is a functional assessment designed to measure the muscular endurance of the elbow extensors. In this test, the participant is seated or standing and holds a 1 kg weight in their hand. The arm starts in a flexed position with the elbow bent at approximately 90 degrees. The participant then extends the elbow fully and returns to the starting flexed position, repeating this movement as many times as possible within a 30-second period. The number of complete flexion-extension cycles performed within the timeframe is counted and recorded. The primary variable measured in this test is the number of repetitions completed within the 30-second timeframe. This is a quantitative variable representing the muscular endurance of the elbow extensors. Specifically, it is a discrete variable since it counts the number of distinct repetitions performed.
Change in lower extremity strength measured with the 30 Seconds Sit-to-Stand Test, at baseline and at the end of the program. | 9 weeks
  The test is particularly useful for evaluating older adults but can also be applied to younger populations and athletes. The primary objective of the 30CST is to measure the number of times a participant can transition from a seated to a standing position and back to seated within a 30-second period. This test is part of the Fullerton Functional Fitness Test Battery and was developed to overcome the limitations of the five or ten repetition sit-to-stand tests, which often exhibit a floor effect in older adults. The measurement that it is used in this test is a quantitative discrete variable.
Change in C-reactive protein measured in blood samples, at baseline and at the end of the program. | 9 weeks
  The C-reactive protein (CRP) is a blood test that measures the level of the CRP protein in the blood. CRP is produced by the liver in response to inflammation in the body. The change in CRP levels measured from blood samples can be used to assess the degree of inflammation and monitor the effectiveness of treatment. It is measured in Milligrams per deciliter (mg/dL).
Change in Neutrophil-to-Lymphocyte Ratio in blood samples, at baseline and at the end of the program. | 8 months
  The neutrophil-to-lymphocyte ratio (NLR) is a simple calculation obtained by dividing the absolute neutrophil count by the absolute lymphocyte count from a complete blood count with differential. It serves as an indicator of systemic inflammation, with higher values reflecting an increased inflammatory state, it is measured in mm³.
Residual cancer burden score after neoadjuvant treatment. | 8 months
  The RCB score is calculated based on several pathological parameters, including the size of the residual tumor, the percentage of the tumor that is invasive, the extent of lymph node involvement, and the size of the largest nodal metastasis. The RCB score is a continuous index that categorizes patients into four classes based on the level of residual disease: RCB-0: Pathologic complete response (no residual invasive cancer), RCB-I: Minimal residual disease, RCB-II: Moderate residual disease and RCB-III: Extensive residual disease.
Pathological complete response measured after neoadjuvant chemotherapy | 8 months
  Pathological complete response is a critical endpoint in the evaluation of neoadjuvant chemotherapy for breast cancer. It is defined as the absence of residual invasive cancer in the breast and axillary lymph nodes following treatment. This response is considered a surrogate marker for long-term outcomes such as overall survival and event-free survival. Is a binary outcome variable that indicates whether a patient achieved complete eradication of invasive cancer in the breast and lymph nodes after receiving neoadjuvant chemotherapy for breast cancer.
Change in lipid profile measured by Low Density Lipoprotein on blood sample, at baseline and at the end of the program. | 9 weeks
  Low-Density Lipoprotein (LDL) measurement in a blood sample using the enzymatic method will be performed. This method involves several enzymatic reactions to quantify the levels of cholesterol and triglycerides. The Friedewald formula is then used to calculate LDL cholesterol (LDL-C) when direct measurement isn't feasible. The formula is:
  LDL-C=Total Cholesterol-HDL Cholesterol-(Triglycerides5)LDL-C=Total Cholesterol-HDL Cholesterol-(5Triglycerides) Here, Total Cholesterol, HDL Cholesterol, and Triglycerides are measured enzymatically. The triglyceride value is divided by 5 to estimate Very Low-Density Lipoprotein (VLDL) cholesterol. The units for these measurements are typically milligrams per deciliter (mg/dL).
  In this context, the variable type for LDL cholesterol is continuous, as it can take on any value within a range and is measured on a continuous scale. The unit of measurement is Milligrams per deciliter (mg/dL).
Change in lipid profile measured by High Density Lipoprotein on blood sample, at baseline and at the end of the program. | 9 weeks
  HDL cholesterol in blood is measured using the enzymatic method, which involves specific enzymatic reactions. A blood sample is prepared and treated to isolate HDL cholesterol. Enzymes such as cholesterol esterase hydrolyze HDL cholesterol esters into free cholesterol. Cholesterol oxidase then oxidizes the free cholesterol, producing hydrogen peroxide (H₂O₂). In the presence of peroxidase, H₂O₂ reacts with a chromogenic substrate to produce a colored compound. The intensity of this color, measured spectrophotometrically, is directly proportional to the HDL cholesterol concentration. A calibration curve, generated using known HDL cholesterol standards, allows determination of the sample's HDL cholesterol concentration by comparing color intensity. The unit of measurement is Milligrams per deciliter (mg/dL).
Change in lipid profile measured by Red Blood Cell membrane Fatty Acid w3 on blood sample, at baseline and at the end of the program. | 9 weeks
  The change in ω-3 fatty acids in the red blood cell (RBC) membrane is measured to assess alterations in lipid profiles. A blood sample is collected, and RBCs are isolated. Lipids are extracted from the RBC membrane using solvents, and the extracted lipids are converted to fatty acid methyl esters (FAMEs). These FAMEs are analyzed using gas chromatography, which separates and quantifies individual fatty acids. The ω-3 fatty acids are expressed as a percentage of total fatty acids.
Change in lipid profile measured by Red Blood Cell membrane Fatty Acid w6 on blood sample, at baseline and at the end of the program. | 9 weeks
  The change in ω-6 fatty acids in the red blood cell (RBC) membrane is measured to evaluate alterations in lipid profiles. A blood sample is collected, and RBCs are isolated. Lipids are extracted from the RBC membrane using solvents, and these lipids are converted to fatty acid methyl esters (FAMEs). The FAMEs are analyzed using gas chromatography, which separates and quantifies individual fatty acids. The ω-6 fatty acids are expressed as a percentage of total fatty acids.
Change in lipid profile measured by the 24-hour dietary recall questionnaire, at baseline and at the end of the program. | 9 weeks
  This instrument provides comprehensive, quantitative information on individual diets by querying respondents about the type and quantity of all food and beverages consumed in the previous 24 hours. This method yields data that can be analyzed to assess dietary patterns, food groups, or nutrient intake. To analyze the nutrient content, the food data must be matched with nutrient information from a food composition database, allowing for the estimation of mean intakes of foods and nutrients.

CONTACTS AND LOCATIONS:
Overall Officials: Viviana Montecinos, Professor, Study Director — Pontifica Universidad católica de Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ramirez K, Acevedo F, Herrera ME, Ibanez C, Sanchez C. [Physical activity and breast cancer]. Rev Med Chil. 2017 Jan;145(1):75-84. doi: 10.4067/S0034-98872017000100011. Spanish. PMID 28393973
- [Background] Acevedo F, Walbaum B, Medina L, Merino T, Camus M, Puschel K, Ramirez K, Manzor M, Veglia P, Martinez R, Guerra C, Navarro M, Bauerle C, Dominguez F, Sanchez C. Clinical characteristics, risk factors, and outcomes in Chilean triple negative breast cancer patients: a real-world study. Breast Cancer Res Treat. 2023 Jan;197(2):449-459. doi: 10.1007/s10549-022-06814-x. Epub 2022 Nov 21. PMID 36414796
- [Background] Valenzuela R, Walbaum B, Farias C, Acevedo F, Vargas C, Bennett JT, Bravo ML, Pinto MP, Medina L, Merino T, Ibanez C, Parada A, Sanchez C. High linoleic acid levels in red blood cells predict a poor response to neoadjuvant chemotherapy in human epidermal growth factor receptor type 2-positive breast cancer patients. Nutrition. 2024 May;121:112357. doi: 10.1016/j.nut.2024.112357. Epub 2024 Jan 9. PMID 38430738
- [Derived] Montt-Blanchard D, Ramirez-Parada K, Montecinos V. Home-based patient-centered physical activity program for quality of life preservation during neoadjuvant chemotherapy in breast cancer: the AURORA randomized controlled trial protocol. Trials. 2026 Jan 7;27(1):12. doi: 10.1186/s13063-025-09301-y. PMID 41501916